CLINICAL TRIAL: NCT05207969
Title: Efficacy of the Act of Urination to Relief the Pain During Flexible Cystoscopy Procedure.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Munawwar Bin Mohd Adnan, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUSMKK
Record Dates: First submitted 2021-06-29; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Hematuria; Bladder Ca; Bladder Stone; Urologic Diseases
MeSH Terms: conditions — Hematuria; Urinary Bladder Neoplasms; Urinary Bladder Calculi; Urologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Cystoscopy procedure will be done based on cystoscopy protocol. During scope procedure patient will not giving instruction to urinate during the procedure.
- Experimental Arm (Experimental): Cystoscopy procedure will be done based on cystoscopy protocol. During scope procedure, patient will be ask to urinate and this will lead to contraction of urinary bladder and relaxation of external urethral sphincter. Scope will then pass through external urethral sphinter and go to the urinary bladder
  Interventions: Procedure: Instruction to urinate

INTERVENTIONS:
Procedure: Instruction to urinate — Cystoscopy procedure will be done based on cystoscopy protocol. During scope procedure, patient will be ask to urinate and this will lead to contraction of urinary bladder and relaxation of external urethral sphincter. Scope will then pass through external urethral sphinter and go to the urinary bladder
  Other Names: voiding instruction
  Arms: Experimental Arm

SUMMARY:
This research is about modification during routine cystoscopy (scope in the bladder) procedure [ experimental research ]. The goal of the study is to evaluate patient experience with cystoscopy by using procedural modification to reduce pain perception. The investigator aim for quality improvement of the current methods of cystoscopy to achieve a better patient experience.

DETAILED DESCRIPTION:
Study Area

-Department of Urology, Hospital Universiti Sains Malaysia.

Study population. -Patient who is required for flexible cystoscopy procedure attending Urology Unit in Hospital USM

Participants

Inclusion Criteria :

• Adult (>18 years old)

Exclusion criteria:

* Analgesic use within 24hours
* History of stricture ,urinary tract infection, existing urethral pain
* Secondary procedure(example stent, stone removal, fulguration)

Withdrawal Criteria

* Change of mind
* Found to be outside the parameters of inclusion criteria, and inside the parameters of exclusion criteria
* Breach of Protocol

ELIGIBILITY:
Inclusion Criteria:

* age more 18 years old

Exclusion Criteria:

* Analgesic use within 24hours
* History of stricture ,urinary tract infection, existing urethral pain
* Secondary procedure(exp stent, stone removal, fulguration)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
1)To determine the efficacy of the act of urination in reducing patient urethral pain during flexible cystoscopy procedure. | During cystoscopy procedure
  To determine the efficacy of the act of urination , we will use visual analogue score (VAS) , subjective assessment for assessing the patient pain score.

SECONDARY OUTCOMES:
2)To determine the association between the act of urination with relaxation of external urethral sphincter during flexible cystoscopy procedure. | During cystoscopy procedure
  We will use electromyography (EMG) as objective assessent to determine association between act of urination and relaxation of external urethral sphinter.

CONTACTS AND LOCATIONS:
Overall Officials: MUNAWWAR BIN ADNAN DR, MD, Principal Investigator — HUSM
Locations (1):
- Hospital University Sains Malaysia, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No